CLINICAL TRIAL: NCT06763913
Title: taVNS Reduces Postoperative Pain and Complications in Patients With Gastric and Intestinal Tumors: A Randomized, Double-Blind, Parallel-Controlled Trial
Brief Title: taVNS Reduces Postoperative Pain and Complications in Patients With Gastric and Intestinal Tumors
Acronym: taVNS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-1127
Record Dates: First submitted 2024-12-15; First posted 2025-01-08 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2024-12

CONDITIONS: taVNS; Gastrointestinal Tumor Surgery; Visual Analogue Scale; Complications
Keywords: taVNS; Perioperative period; Visual Analogue Scale; complications

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- taVNS (Experimental): Set the pulse width to 200 microseconds, frequency to 30 Hz, and start the current at 10 mA. Gradually increase the current until the patient reaches their pain tolerance threshold, and cap it at 50 mA.
  Interventions: Device: taVNS
- sham taVNS (Sham Comparator): Set the pulse width to 200 microseconds, frequency to 1 Hz, current to 10 mA and gradually increase it to the patient's pain tolerance threshold, capped at 50 mA.
  Interventions: Device: sham taVNS

INTERVENTIONS:
Device: taVNS — Set the pulse width to 200 microseconds, frequency to 30 Hz, and start the current at 10 mA. Gradually increase the current until the patient reaches their pain tolerance threshold, and cap it at 50 mA，last for one hour.During the intervention, dynamic ECG monitoring was conducted using an ECG monitor, starting 10 minutes before the stimulation and ending 10 minutes after the stimulation.
  Arms: taVNS
Device: sham taVNS — Set the pulse width to 200 microseconds, frequency to 1 Hz, and start the current at 10 mA. Gradually increase the current until the patient reaches their pain tolerance threshold, and cap it at 50 mA，last for one hour.During the intervention, dynamic ECG monitoring was conducted using an ECG monitor, starting 10 minutes before the stimulation and ending 10 minutes after the stimulation.
  Arms: sham taVNS

SUMMARY:
Postoperative acute pain control in patients with gastrointestinal tumors is not satisfactory, and surgical complications including gastrointestinal dysfunction, gastrointestinal fistula, abdominal and gastrointestinal hemorrhage, peritonitis and abscess, are still important factors affecting surgical outcomes, postoperative recovery, hospital stay, and even perioperative mortality. The application of taVNS during the perioperative period can enhance or preserve vagal nerve function, which may protect important organ functions through multiple pathways such as alleviating pain and inflammatory responses caused by surgical trauma, improving gastrointestinal function, enhancing cardiovascular regulation, reducing postoperative nausea and vomiting, and accelerating postoperative recovery, thereby reducing postoperative complications and mortality.

DETAILED DESCRIPTION:
Subjects who met the inclusion criteria were enrolled in the clinical trial and received 2 interventions at the following times: the day before surgery, and the afternoon of the 1st day postoperatively (15:00-17:00), a total of 2 times. The intervention implementers used vagus nerve stimulation equipment to place electrodes in the tragus area of the outer ear of the subjects in the experimental group (taVNS group). The control group (sham stimulation group) was set to have a pulse width of 200 μs, a frequency of 1 Hz, and an initial current of 10 mA, which was gradually increased to the pain tolerance threshold of the subject, capped at 50 mA，last for one hour. The VAS scores before and after stimulation for 10 minutes were recorded.

2) ECG monitoring: Both groups were monitored with a dynamic ECG monitor during the intervention period, starting 10 minutes before stimulation and ending 10 minutes after stimulation. The SDNN (Standard Deviation of NN intervals) of the sinus rhythm was measured before and after stimulation for 10 minutes. A uniform standard was used for anesthesia induction and maintenance during surgery, and all patients used the same patient-controlled intravenous analgesia (PCIA) plan.

ELIGIBILITY:
Inclusion Criteria:

Age 18-80 years, BMI 18-30 kg/m², ASA Ⅱ-Ⅲ, elective laparoscopic gastric or intestinal tumor surgery, expected surgical duration ≥2 hours, patient understands study content and signs informed consent form.

Exclusion Criteria:

Kidney replacement therapy, treatment for arrhythmias requiring treatment, dementia, severe bradycardia, orthostatic tachycardia syndrome, neuro-muscular disorders, auricular dermatitis, planned post-operative transfer to ICU

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Difference in VAS Score on Postoperative Day 1 | before and after each stimulus for 10 minutes
  Difference in VAS Score on Postoperative Day 1

SECONDARY OUTCOMES:
The QoR-15 scale scores on the 1st and 3rd days after surgery | 1 day before the operation and the third day after the operation
  The QoR-15 scale scores on the 1st and 3rd days after surgery
Postoperative Complication Rate | 1 day before being discharged from the hospital
  Postoperative in-hospital complication rate
The time of the first postoperative anal exhaust | On the third day after the operation
  The time of the first postoperative anal exhaust
The effective number of pain relief pump presses | One day before being discharged from the hospital
  The effective number of pain relief pump presses
Postoperative Salvage Analgesic Consumption of Opioid Equivalents | One day before being discharged from the hospital
  Postoperative Salvage Analgesic Consumption of Opioid Equivalents
Length of hospital stay | One day before being discharged from the hospital
  Length of hospital stay
Standard Deviation of NN intervals | 10 minutes before and after each stimulus
  10 minutes before and after each stimulus
Root Mean Square of the Successive Differences | 10 minutes before and after each stimulus
  10 minutes before and after each stimulus

CONTACTS AND LOCATIONS:
Locations (1):
- Second affiliated Hospital School of Medicine, Hangzhou, Zhejiang, China